CLINICAL TRIAL: NCT05849077
Title: Optimization of Saturation Targets And Resuscitation (OptiSTART): Multicenter Randomized Controlled Trial
Brief Title: Optimization of Saturation Targets And Resuscitation Trial (OptiSTART)
Acronym: OptiSTART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Oklahoma (Other); North Central Baptist Hospital (Unknown); Sharp Mary Birch Hospital for Women & Newborns (Other); The Woman's Hospital of Texas (Other); Baylor College of Medicine (Other); University of Florida Health (Other); University of Pittsburgh Medical Center (Other); University of Pittsburgh (Other); University of Utah (Other); Primary Children's Hospital (Other); Methodist Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Vishal Kapadia, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2022-0441
Record Dates: First submitted 2023-04-21; First posted 2023-05-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Premature Infants; Bronchopulmonary Dysplasia; Intraventricular Hemorrhage; Neurodevelopmental Outcomes
Keywords: neonatal resuscitation; oxygen
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sat75 (Experimental): FiO2 will be titrated every 30 seconds by 0.2-0.3 to achieve target SpO2 that approximates the 75th percentile SpO2 observed in healthy term newborns. Percentiles are roughly based on Dawson reference curves of healthy term infants after birth.
  Interventions: Other: Sat75
- Sat50 (Active Comparator): FiO2 will be titrated every 30 seconds by 0.1-0.2 to achieve NRP recommended target SpO2 which approximates the 50th percentile SpO2 observed in healthy term newborns. Percentiles are roughly based on Dawson reference curves of healthy term infants after birth.
  Interventions: Other: Sat50

INTERVENTIONS:
Other: Sat75 — As per the current NRP guidelines, resuscitation will be initiated with 0.3 FiO2. FiO2 will be titrated every 30 seconds by 0.2-0.3 to achieve target SpO2 that approximates the 75th percentile SpO2 observed in healthy term newborns. Percentiles are roughly based on Dawson reference curves of healthy term infants after birth. Apart from the randomly assigned target SpO2, resuscitation will follow the current NRP guidelines. Following NICU admission, all care decisions, including ventilator management, will be at the discretion of the clinical team.
  Arms: Sat75
Other: Sat50 — As per the current NRP guidelines, resuscitation will be initiated with 0.3 FiO2. FiO2 will be titrated every 30 seconds by 0.1-0.2 to achieve target SpO2 that approximates the 50th percentile SpO2 observed in healthy term newborns. Percentiles are roughly based on Dawson reference curves of healthy term infants after birth. Apart from the randomly assigned target SpO2, resuscitation will follow the current NRP guidelines. Following NICU admission, all care decisions, including ventilator management, will be at the discretion of the clinical team.
  Arms: Sat50

SUMMARY:
This study is designed to answer one of the fundamental gaps in knowledge in the resuscitation of preterm infants at birth: What is the optimal target oxygen saturation (SpO2) range that increases survival without long-term morbidities? Oxygen (O2) is routinely used for the stabilization of preterm infants in the delivery room (DR), but its use is linked with mortality and several morbidities including bronchopulmonary dysplasia (BPD). To balance the need to give sufficient O2 to correct hypoxia and avoid excess O2, the neonatal resuscitation program (NRP) recommends initiating preterm resuscitation with low (≤ 30%) inspired O2 concentration (FiO2) and subsequent titration to achieve a specified target SpO2 range. These SpO2 targets are based on approximated 50th percentile SpO2 (Sat50) observed in healthy term infants. However, the optimal SpO2 targets remain undefined in the preterm infants. Recent data suggest that the current SpO2 targets (Sat50) may be too low. The investigators plan to conduct a multicenter RCT of Sat75 versus Sat50 powered for survival without BPD. The investigators will randomize 700 infants, 23 0/7- 30 6/7 weeks' GA, to 75th percentile SpO2 goals (Sat75, Intervention) or 50th percentile SpO2 goals (Sat50, control). Except for the SpO2 targets, all resuscitations will follow NRP guidelines including an initial FiO2 of 0.3. In Aim 1, the investigators will determine whether targeting Sat75 compared to Sat50 increases survival without lung disease (BPD). In addition, the investigators will compare the rates of other major morbidities such as IVH. In Aim 2, the investigators will determine whether targeting Sat75 compared to Sat50 increases survival without neurodevelopmental impairment at 2 years of age. In Aim 3, the investigators will determine whether targeting Sat75 compared to Sat50 decreases oxidative stress.

DETAILED DESCRIPTION:
Purpose: Oxygen is the most commonly used drug during preterm resuscitation, but its use has been linked to mortality and several morbidities such as bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH), and retinopathy of prematurity (ROP).Preterm infants at birth are more vulnerable to oxygen toxicity caused by exposure to high concentrations of oxygen during resuscitation, but are also equally vulnerable to the adverse effects of suboptimal oxygen use in the delivery room. To balance the need to give sufficient O2 to correct hypoxia and to avoid excess O2, the NRP recommends initiating preterm resuscitation with low FiO2 (≤ 0.3) and subsequent titration to achieve specified target O2 saturations (SpO2). These SpO2 targets (Sat50) are based on approximated 50th percentile SpO2 values of minute per minute pre-ductal SpO2 observed in healthy term newborns who were born vaginally at sea level, breathing spontaneously and did not need any oxygen at birth. Current SpO2 targets are based on expert opinion. In the absence of studies comparing different SpO2 targets, Sat50 was selected by experts at the International Liaison Committee On Resuscitation (ILCOR) and NRP to balance the need for O2 supplementation and avoid excess O2 exposure. Ranges were adjusted by NRP so that they could be memorized easily. However, a recently published study suggested that the currently recommended Sat50 targets are lower than 50th percentile SpO2 values for term infants who undergo delayed cord clamping. Recent studies suggest that the currently recommended Sat50 SpO2 targets may be too low to promote an adequate drop in pulmonary vascular resistance in preterm infants and may be harmful. Recent studies raise concern that the Sat50 strategy may be associated with poorer breathing efforts, higher IVH and higher mortality. The majority of research in O2 use during preterm resuscitation has focused on the starting FiO2, while SpO2 targets have received very little attention. The investigators propose a paradigm shift by changing the research focus to determine the optimal target SpO2 range instead of the initial FiO2. The investigators propose a novel O2 strategy where resuscitation is initiated with 0.3 FiO2 and is titrated every 30 seconds to meet target SpO2 roughly based on the 75th percentile of Dawson curves (Sat75) compared to the 50th percentile of Dawson curves (Sat50). Preliminary data from principal investigator's NICHD K23 funded pilot RCT of 75 preterm infants <31 weeks' gestational age (GA) demonstrated that infants randomized to 75th percentile SpO2 goals (Sat75) had a lower incidence of SpO2 <80% at five minutes and lower duration of bradycardia and PPV in the DR compared to infants randomized to 50th percentile SpO2 goals (Sat50). Although not powered for this analysis, Sat75 infants had less pulmonary hypertension and higher survival without BPD. The investigators hypothesize that the Sat75 strategy results in better pulmonary transition, less time with low SpO2 and lower oxidative stress resulting in a lower incidence of neonatal morbidities such as BPD, IVH, ROP and higher survival without BPD.

Hypothesis: The primary hypothesis is that delivery room resuscitation of preterm infants < 31 weeks' GA with Sat75 targets compared to Sat50 targets will result in increased survival without BPD at 36 weeks' postmenstrual age (PMA).

Study design: A prospective multicenter randomized controlled trial of Sat75 versus Sat50 will be conducted. As per the current NRP guidelines, resuscitation will be initiated with 0.3 FiO2 in both intervention and control groups. The study intervention is the Sat75 where FiO2 will be titrated every 30 seconds by 0.1-0.2 to achieve target SpO2 that approximates the 75th percentile SpO2 observed in healthy term newborns. The control group is the Sat50 where FiO2 will be titrated by 0.2-0.3 every 30 seconds to achieve the NRP recommended target SpO2 which approximates the 50th percentile SpO2 observed in healthy term newborns. In the rare event, where chest compressions are needed during delivery room resuscitation, the FiO2 will be increased to 1.0 as per current NRP guidelines. Once the heart rate (HR) is stabilized, the FiO2 will be reduced to meet the target SpO2. Apart from the randomly assigned target SpO2, resuscitation will follow current NRP guidelines. Assignment to the Sat75 or Sat50 group will use a 1:1 allocation ratio and stratification by GA: 23 0/7 to 27 6/7 weeks and 28 0/7 to 30 6/7 weeks. Demographics, perinatal variables, resuscitation characteristics and neonatal morbidity-mortality data and data of Neurodevelopmental follow-up at around 2 years of age will be electronically recorded using the web-based data entry system developed by the Data Coordinating Center.

Analysis plan: An intention to treat analysis of all randomized infants who received study intervention and have a post-randomization study measurement will be conducted. Baseline characteristics of the newborns will be compared between treatment groups. Descriptive statistics such as mean, SD, median, and range will be used to summarize continuous variables in each study group; frequencies and percentages will be presented for categorical variables. The groups will be formally compared using Student's t-tests and Wilcoxon rank-sum tests, as appropriate, for continuous variables. The chi-square test of association and Fisher's exact test will be used for categorical variables as appropriate.

The primary analysis will be based on the chi-square test of association. Rates of survival without BPD will be presented with 95% confidence intervals. Multivariable logistic regression models (for odds ratios), or modified Poisson regression models with robust standard errors (for risk ratios), will be used to adjust for any imbalanced baseline characteristics. Any characteristics identified as being imbalanced at baseline will be considered as covariates. The primary analysis plan assumes that the intra-class correlation among infants of multiple gestations will be negligible. As sensitivity analyses, generalized estimating equations with robust standard errors will be used to account for clustering effects within siblings. Statistical analysis will be performed with SAS software version 9.4 (SAS Institute, Cary NC). A two-sided 0.05 level of significance will be used and no interim analysis is planned. Data collection protocols will be implemented to minimize missing data. The investigators will conduct 'Per Protocol' analysis and 'As Treated' analysis strictly as secondary analyses to evaluate the impact of time spent outside the group target SpO2 on clinical outcomes. Further, the investigators will conduct pre-planned analyses to examine possible site by testing site by treatment interactions.

ELIGIBILITY:
Inclusion Criteria:

-Neonates with OB gestational age 22-30 weeks

Exclusion Criteria:

* Prenatally diagnosed cyanotic congenital heart disease
* Prenatally diagnosed congenital diaphragmatic hernia
* Parents request no resuscitation
* If preductal saturations can not be measured by 3 minutes after pulse oximeter sensor is applied to the newborn

Ages: 0 Minutes to 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Survival without BPD | 36 weeks Postmenstrual Age
  The primary outcome for this trial is survival without BPD at 36 weeks' PMA. Both components, death and BPD, will also be reported separately. Neonatal mortality during the NICU stay, the postnatal day at the time of mortality and the primary cause of mortality will be recorded. BPD will be defined as the need for any form of positive airway pressure support or supplemental O2 at 36 weeks' PMA.BPD will be graded as mild, moderate and severe as per the NICHD consensus definition. All eligible infants will undergo room air challenge at 36 weeks' PMA for the physiologic definition of BPD.

SECONDARY OUTCOMES:
Bronchopulmonary Dysplasia | 36 weeks PMA, 40 weeks PMA and at Discharge
  BPD will be defined as the need for any form of positive airway pressure support or supplemental O2 at 36 weeks' PMA.BPD will be graded as mild, moderate and severe as per the NICHD consensus definition. All eligible infants will undergo room air challenge at 36 weeks' PMA for the physiologic definition of BPD. In addition, BPD by Jensen Criteria will also be used as a secondary outcome. Respiratory support at 40 weeks PMA and at discharge will also be collected
Oxygen saturations in the delivery room | First 15 minutes after birth
  High resolution SpO2 data with 2 second frequency from pulse oximeter will be collected. Average Spo2 value every 30 seconds will be plotted. The investigators will also calculate time spent in the desired target, above the target or below the target.
SpO2<80% at 5 minutes after birth | First 5 minutes after birth
  SpO2<80% at 5 minutes after birth
Delivery Room Intubation | Up to first 30 minutes after birth
  The investigators will record if the newborn was intubated in the delivery room
Receipt of chest compressions and epinephrine | Up to first 30 minutes after birth
  In the rare event of the need for full CPR, data will be abstracted from the DR code documentation. FiO2 will be adjusted to 1.0 until return of spontaneous circulation and then titrated to achieve the randomized target SpO2.
Severe Intraventricular hemorrhage | From date of randomization until the date of first documented diagnosis or date of death from any cause or date of discharge, whichever came first, assessed up to 12 months
  Severe Intraventricular hemorrhage
Severe Retinopathy of Prematurity | From date of randomization until the date of first documented diagnosis or date of death from any cause or date of discharge, whichever came first, assessed up to 12 months
  Severe Retinopathy of Prematurity
Length of hospitalization | From date of randomization until the date of first documented diagnosis or date of death from any cause or date of discharge, whichever came first, assessed up to 12 months
  Length of hospitalization
Necrotizing Enterocolitis (NEC) | From date of randomization until the date of first documented diagnosis or date of death from any cause or date of discharge, whichever came first, assessed up to 12 months
  Necrotizing enterocolitis will be defined ≥ Stage 2 based on the modified Bell criteria.
Neurodevelopmental Impairment (NDI) | From date of randomization until the date of first documented diagnosis or date of death from any cause or date of discharge, whichever came first, assessed up to 36 months
  Moderate to severe neurodevelopmental impairment will be defined as Bayley III Cognitive <85, Bayley III Motor <85, gross motor functional classification system (GMFCS) 2 or greater, or bilateral "blind" despite corrective lenses or bilateral no functional hearing with or without amplification
Oxidative Stress | from time of randomization to the first 24 hours after birth
  8-Isoprostanes and 8-OHdG will be measured in serum and urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Kapadia, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per NICHD requirements (National Institute of Child Health and Human Development). Researchers can email the PI for more information at vishal.kapadia@utsouthwestern.edu
Supporting Information: CSR
Time Frame: After the completion of data analysis and manuscript publication.
Access Criteria: An archived dataset with documentation will be made available for additional uses by outside investigators, in collaboration with the study investigators.